CLINICAL TRIAL: NCT05078060
Title: Enhanced Passive Safety Surveillance of VaxigripTetra® (Quadrivalent Inactivated Split Virion Influenza Vaccine, Intramuscular Route) and Efluelda® (Quadrivalent Inactivated Split Virion Influenza Vaccine, Intramuscular Route) Vaccines in Europe During the Influenza Season 2021/22.
Brief Title: Safety Surveillance of VaxigripTetra® and Efluelda® Influenza Vaccines in Europe During the Influenza Season 2021/22
Status: Completed | Type: Observational
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Other Study IDs: FLU00170
Record Dates: First submitted 2021-10-01; First posted 2021-10-14 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03-03

CONDITIONS: Influenza (Healthy Volunteers)
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- VaxigripTetra®: Participant vaccinated with VaxigripTetra® as per routine clinical practice
  Interventions: Biological: Quadrivalent Influenza Vaccine
- Efluelda®: Participant vaccinated with Efluelda® as per routine clinical practice
  Interventions: Biological: High-Dose Quadrivalent Influenza Vaccine

INTERVENTIONS:
Biological: Quadrivalent Influenza Vaccine — Intramuscular or subcutaneous administration
  Other Names: VaxigripTetra®
  Groups: VaxigripTetra®
Biological: High-Dose Quadrivalent Influenza Vaccine — Intramuscular administration
  Other Names: Efluelda®
  Groups: Efluelda®

SUMMARY:
The primary objective of the study is to estimate the reporting rate of suspected Adverse Drug Reactions (ADRs) occurring within 7 days following routine vaccination with VaxigripTetra® and Efluelda®, respectively, during the Northern Hemisphere (NH) influenza season 2021/22.

The secondary objectives of the study are:

* To estimate the reporting rates of suspected ADRs occurring within 7 days following routine vaccination with VaxigripTetra® according to the pre-defined age groups.
* To estimate the reporting rates of serious suspected ADRs after vaccination with VaxigripTetra®, and Efluelda®, respectively, at any time following vaccination, within the Enhanced Passive Safety Surveillance (EPSS) period.
* To compare vaccinees' reporting rates of suspected ADRs observed during the NH influenza season 2021/22.

DETAILED DESCRIPTION:
Study duration per participant is maximum 2 months.

ELIGIBILITY:
Individuals who approach the site for vaccination and agree to receive a vaccination card will be included and vaccinated with the respective vaccine brand according to the country of their location, recommendations for the individual vaccines as well as national recommendations.

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: VaxigripTetra® will be given to adults (including pregnant women) and children aged 6 months and older in Finland. Efluelda® will be given to adults 60 years of age and older in Germany.
Sampling Method: Non-Probability Sample
Enrollment: 1804 (Actual)
Dates: Start 2021-10-12 (Actual); Primary Completion 2021-12-02 (Actual); Study Completion 2021-12-02 (Actual)

PRIMARY OUTCOMES:
Vaccinees' reporting rate following routine vaccination with VaxigripTetra® and Efluelda® | Within 7 days after vaccination
  The vaccinees' reporting rate is expressed as the percentage of vaccinees who reported at least one suspected ADR among the distributed vaccination cards
ADR reporting rate following routine vaccination with VaxigripTetra® and Efluelda® | Within 7 days after vaccination
  The ADR reporting rate is expressed as the percentage of suspected ADRs among the distributed vaccination cards

SECONDARY OUTCOMES:
ADR reporting rate according to age group | Within 7 days after vaccination
Vaccinees' reporting rate according to age group | Within 7 days after vaccination
Vaccinees' reporting rate of serious suspected ADRs at any time following vaccination within the EPSS period | From vaccination to end of data collection (maximum 2 months following first vaccination)
  Serious suspected ADRs will be collected from vaccination up to the end of data collection. Data collection ends when 1000 vaccination cards have been distributed (per vaccine brand) plus 2 weeks or 2 months following the first vaccination, whichever comes first.
Serious suspected ADR reporting rate at any time following vaccination within the EPSS period | From vaccination to end of data collection (maximum 2 months following first vaccination)
  Serious suspected ADRs will be collected from vaccination up to the end of data collection. Data collection ends when 1000 vaccination cards have been distributed (per vaccine brand) plus 2 weeks or 2 months following the first vaccination, whichever comes first.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (15):
- Finland (5):
  - Investigational Site Number :2-2-002, Helsinki
  - Investigational Site Number :2-2-005, Jyväskylä
  - Investigational Site Number :2-2-004, Kuopio
  - Investigational Site Number :2-2-003, Tampere
  - Investigational Site Number :2-2-011, Turku
- Germany (10):
  - Investigational Site Number :2760005, Blankenhain
  - Investigational Site Number :2760008, Bochum
  - Investigational Site Number :2760001, Donaueschingen
  - Investigational Site Number :2760011, Düsseldorf
  - Investigational Site Number :2760007, Frankfurt am Main
  - Investigational Site Number :2760002, Fulda
  - Investigational Site Number :2760003, Grafenrheinfeld
  - Investigational Site Number :2760004, Haar
  - Investigational Site Number :2760006, Hamburg
  - Investigational Site Number :2760009, Wendelstein

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Background] Gandhi-Banga S, Wague S, Shrestha A, Syrkina O, Talanova O, Nissila M, Stuff K, Monfredo C. Enhanced passive safety surveillance of high-dose and standard-dose quadrivalent inactivated split-virion influenza vaccines in Germany and Finland during the influenza season 2021/22. Influenza Other Respir Viruses. 2023 Jan;17(1):e13071. doi: 10.1111/irv.13071. Epub 2022 Nov 29. PMID 36448240